CLINICAL TRIAL: NCT01058200
Title: Assess the Risk-benefit Balance of the New Vacuum Assisted-delivery Device "iCUP" Versus the Reference Vacuum. Multicenter Prospective Randomized Controlled Study
Brief Title: a Randomized Multicenter Trial Comparing Vacuum Assisted Delivery With the New Device "iCUP" Versus the Reference Cup.
Acronym: ICUP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurCIC, Dr Véronique EQUY, University Hospital, Grenoble., University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 07 23
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Vacuum Extraction, Obstetrical; Randomized Controlled Trials; Failures, Medical Device; Maternal Lesions; Neonatal Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vacuum extractor 'iCUP' (Active Comparator): new vacuum extractor: sterile disposable plastic cup
  Interventions: Device: iCup
- reference vacuum extractor (Sham Comparator): reference cup of the obstetrical ward: metallic cup
  Interventions: Device: reference cup

INTERVENTIONS:
Device: iCup — new vacuum extractor: sterile disposable plastic cup
  Arms: vacuum extractor 'iCUP'
Device: reference cup — reference cup of the obstetrical ward: metallic cup
  Arms: reference vacuum extractor

SUMMARY:
The hypothesis is that the new vacuum assisted delivery device iCup is more effective than the reference cup, in terms of maternal and newborn morbidities and functioning

DETAILED DESCRIPTION:
Currently, instrumental extractions are used in about 10% to 15% of the 860 000 annual deliveries in France and the use of vacuum extractors increases from year to year. In addition to sterilizable vacuum extractors several different types of vacuum extractor have been developed, in particular the single use Kiwi cup or the so-called 'soft' cup extractors. However, studies evaluating these new cups have not shown their superiority in comparison to the conventional metallic vacuum extractor.

Accordingly, it is legitimate to assess the new vacuum extractor iCup, an innovative "mix" of metallic cup and 'soft' cups that should combine the advantages of both; and to compare the iCup vacuum extractor with the sterilizable metallic cup extractor, the most effective vacuum extractors available to date.

ELIGIBILITY:
Inclusion Criteria:

* maternal age between 18 and 45 years old
* singleton delivery after 37 weeks, in cephalic presentation,
* indication of vacuum extraction,
* affiliation to the french social security system or equivalent

Exclusion Criteria:

* no informed consent
* singleton delivery before 37 weeks, in non-cephalic presentation,
* patient deprived of freedom

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 668 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Composite outcome: cup detachments (failure=3 detachments), other instrument used, caesarean section, caput succedaneum, cephalohaematoma, maternal perineal lesions. If one of these criteria at least is present, outcome is noted 'failure'; else 'success' | one day

SECONDARY OUTCOMES:
maternal lesions: cervix lesions, postpartum haemorrhage | 28 days maximum
neonatal lesions: minor scalp injuries, Apgar score < 7, pH < 7.20, anaemia, jaundice, transfer | 28 days maximum
medico-economic criteria: cost-effectiveness analysis of the studied medical devices | 28 days maximum

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Patrick SCHAAL, MD PHD, Principal Investigator — University Hospital, Grenoble
Locations (6):
- France (6):
  - University Hospital, Besançon
  - University Hospital, Caen
  - Hospital, Chambéry
  - University Hospital, Clermont-Ferrand
  - University Hospital, Grenoble
  - University Hospital, Strasbourg

REFERENCES:
- [Background] Chalmers JA, Chalmers I. The obstetric vacuum extractor is the instrument of first choice for operative vaginal delivery. Br J Obstet Gynaecol. 1989 May;96(5):505-6. doi: 10.1111/j.1471-0528.1989.tb03246.x. No abstract available. PMID 2757977
- [Background] Johanson R, Menon V. Soft versus rigid vacuum extractor cups for assisted vaginal delivery. Cochrane Database Syst Rev. 2000;(2):CD000446. doi: 10.1002/14651858.CD000446. PMID 10796203
- [Background] Miksovsky P, Watson WJ. Obstetric vacuum extraction: state of the art in the new millennium. Obstet Gynecol Surv. 2001 Nov;56(11):736-51. doi: 10.1097/00006254-200111000-00025. PMID 11711908
- [Background] Schaal JP, Riethmuller D, Menget A. Extractions instrumentales du fœtus : ventouse obstétricale. Encycl Méd Chir Paris: Elsevier, 2004 (vol Obstétrique)
- [Background] Attilakos G, Sibanda T, Winter C, Johnson N, Draycott T. A randomised controlled trial of a new handheld vacuum extraction device. BJOG. 2005 Nov;112(11):1510-5. doi: 10.1111/j.1471-0528.2005.00729.x. PMID 16225571
- [Background] Vacca A. A randomised controlled trial of a new handheld vacuum extraction device. BJOG. 2006 Apr;113(4):492; author reply 494-5. doi: 10.1111/j.1471-0528.2006.00903.x. No abstract available. PMID 16553663
- [Background] Groom KM, Jones BA, Miller N, Paterson-Brown S. A prospective randomised controlled trial of the Kiwi Omnicup versus conventional ventouse cups for vacuum-assisted vaginal delivery. BJOG. 2006 Feb;113(2):183-9. doi: 10.1111/j.1471-0528.2005.00834.x. PMID 16411996
- [Background] Schaal JP, Equy V, Hoffman P. [Comparison vacuum extractor versus forceps]. J Gynecol Obstet Biol Reprod (Paris). 2008 Dec;37 Suppl 8:S231-43. doi: 10.1016/S0368-2315(08)74761-6. French. PMID 19268200
- [Background] Riethmuller D, Ramanah R, Maillet R, Schaal JP. [Vacuum extractors: description, mechanics, indications and contra-indications]. J Gynecol Obstet Biol Reprod (Paris). 2008 Dec;37 Suppl 8:S210-21. doi: 10.1016/S0368-2315(08)74759-8. French. PMID 19268198
- [Derived] Verma GL, Spalding JJ, Wilkinson MD, Hofmeyr GJ, Vannevel V, O'Mahony F. Instruments for assisted vaginal birth. Cochrane Database Syst Rev. 2021 Sep 24;9(9):CD005455. doi: 10.1002/14651858.CD005455.pub3. PMID 34559884
- [Derived] Equy V, David-Tchouda S, Dreyfus M, Riethmuller D, Vendittelli F, Cabaud V, Langer B, Margier J, Bosson JL, Schaal JP. Clinical impact of the disposable ventouse iCup(R) versus a metallic vacuum cup: a multicenter randomized controlled trial. BMC Pregnancy Childbirth. 2015 Dec 15;15:332. doi: 10.1186/s12884-015-0771-1. PMID 26666981